CLINICAL TRIAL: NCT03829800
Title: Effect of the Intake of Specific Formulas for Diabetes With Sucromalt and Isomaltulose on the Glycemic Index, Insulin, Glucagon-like Peptide-1, Gastric Inhibitory Peptide Levels and Subjective Appetite in Subjects With Type 2 Diabetes
Brief Title: Formulas for Diabetes With Sucromalt & Isomaltulose on Glycemic Index, Hormones & Subjective Appetite in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad del Zulia (Other)
Responsible Party: Principal Investigator, Daniel J Aparicio Camargo, Principal Investigator, Universidad del Zulia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 1001092016
Record Dates: First submitted 2019-01-28; First posted 2019-02-04 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Glycemic Index; Insulin; Incretins; Diabetes Mellitus type 2; Subjective appetite; Nutritional formula
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Participants receive 4 nutritional formulas to evaluate their glycemic index, insulin, GLP-1, GIP levels and subjective appetite
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ensure® Abbott Nutrition (Experimental): A standard nutritional formula not specific for diabetics
  Interventions: Dietary Supplement: Ensure® Abbott Nutrition
- Glucerna® Abbott Nutrition (Experimental): A formula with a patented blend of slow-digesting carbohydrates including resistant maltodextrin and sucromalt
  Interventions: Dietary Supplement: Glucerna® Abbott Nutrition
- Diasip® Nutricia Advanced (Experimental): A formula whose composition has isomaltulose and resistant starch
  Interventions: Dietary Supplement: Diasip® Nutricia Advanced
- Glicolab® (Active Comparator): Glucose solution
  Interventions: Dietary Supplement: Glicolab®

INTERVENTIONS:
Dietary Supplement: Ensure® Abbott Nutrition — Effect of the intake of Ensure® Abbott Nutrition on the glycemic index, insulin, GLP-1, GIP levels and subjective appetite in subjects with type 2 diabetes
  Arms: Ensure® Abbott Nutrition
Dietary Supplement: Glucerna® Abbott Nutrition — Effect of the intake of Glucerna® Abbott Nutrition on the glycemic index, insulin, GLP-1, GIP levels and subjective appetite in subjects with type 2 diabetes
  Arms: Glucerna® Abbott Nutrition
Dietary Supplement: Diasip® Nutricia Advanced — Effect of the intake of Diasip® Nutricia Advanced on the glycemic index, insulin, GLP-1, GIP levels and subjective appetite in subjects with type 2 diabetes
  Arms: Diasip® Nutricia Advanced
Dietary Supplement: Glicolab® — Effect of the intake of Glicolab on the glycemic index, insulin and subjective appetite in subjects with type 2 diabetes
  Arms: Glicolab®

SUMMARY:
Consumption of nutritional supplements with low glycemic carbohydrates induce favorable glycemic responses in subjects with type 2 diabetes. The aim of this study was to compare the effect of the intake of specific formulas for diabetes, with different types of carbohydrates (isomaltulose and sucromaltose) on the glycemic response, release of intestinal peptides and subjective appetite in Type 2 diabetic individuals. In a randomized, double-blind, cross-over study of 4 treatments, 16 subjects (56.60 ± 1.11 years). Fasting blood samples were taking, after that they were given to consume formula or reference product assigned randomly. Subsequently, samples of capillary and venous blood were obtained at times 30, 60, 90, 120 and 180 min, after the start of consumption of the experimental beverage for the measurement of glucose, insulin, gastric inhibitory peptide (GIP) and glucagon-like peptide-1 (GLP-1). The assessment of subjective appetite was measured by Visual Analogue Scale (VAS).

DETAILED DESCRIPTION:
This was a randomized, double-blind, cross-over study of 4 treatments that was conducted according to the Good Clinical Practice Guidelines, with all applicable Food and Drug privacy regulations, and ethical principles based on the Declaration of Helsinki. Participants signed informed consent, approved by the Human Research Ethics Committee of the Endocrine-Metabolic Research Center of the University of Zulia, in Venezuela. All selected subjects attended a first visit, in order to determine if they met the inclusion criteria, those who gathered them, were subjected to four consumption tests to determine the glycemic index (GI) and glycemic load (GL) and 3 consumption tests for the evaluation of subjective appetite. Each treatment or consumption session was carried out on different days.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes
* Demonstrated use of oral hypoglycemic agents (metformin), for at least two months
* BMI of 18.5 kg/m2 to ≤ 35 kg/m2

Exclusion Criteria:

* Type 1 Diabetes
* Diabetic ketoacidosis
* Congestive heart failure
* Gastric, renal or hepatic diseases
* Myocardial infarction
* Stroke
* Subjects with insulin therapy, antibiotic therapy or corticosteroids
* End-stage organ failure
* Individuals with organ transplantation
* Coagulation or bleeding disorder
* Infectious or chronic contagious disease (such as tuberculosis, hepatitis B or C or HIV).

Ages: 51 Years to 63 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline Glycemia at 180 minutes | Minutes after intake of each formula: 0, 30, 60, 90, 120, 150, 180.
  mmol/L
Change from baseline Insulin at 180 minutes | Minutes after intake of each formula: 0, 30, 60, 90, 120, 150, 180.
  milliunits per liter (mU/L)
Glycemic Index (GI) | 180 minutes after intake of each formula
  Low GI (≤ 55), Intermediate (55-69) and High (≥70)
Glycemic Load (GL) | 180 minutes after intake of each formula
  High GL (> 20), Intermediate GL (11-19) and Low GL (<10)
Change from baseline GLP-1 at 180 minutes | Minutes after intake of each formula: 0, 30, 60, 90, 120, 150, 180.
  pmol/L
Change from baseline GIP at 180 minutes | Minutes after intake of each formula: 0, 30, 60, 90, 120, 150, 180.
  pg/mL
Change from baseline Hunger at 180 minutes | Minutes after intake of each formula: 0, 30, 60, 90, 120, 150, 180.
  Visual Analogue Scale (mm)
Change from baseline Fullness at 180 minutes | Minutes after intake of each formula: 0, 30, 60, 90, 120, 150, 180.
  Visual Analogue Scale (mm)
Change from baseline Desire to eat at 180 minutes | Minutes after intake of each formula: 0, 30, 60, 90, 120, 150, 180.
  Visual Analogue Scale (mm)
Change from baseline Prospective food consumption at 180 minutes | Minutes after intake of each formula: 0, 30, 60, 90, 120, 150, 180.
  Visual Analogue Scale (mm)
Change from baseline Subjective appetite at 180 minutes | Minutes after intake of each formula: 0, 30, 60, 90, 120, 150, 180.
  Visual Analogue Scale (mm)

SECONDARY OUTCOMES:
Age | Baseline
  years
Weight | Baseline
  kg
Height | Baseline
  m
Body Mass Index | Baseline
  kg/m^2
Hip Circumference | Baseline
  cm
Total Cholesterol | Baseline
  mg/dl
HDL-C | Baseline
  mg/dl
LDL-C | Baseline
  mg/dl
Triacylglycerides | Baseline
  mg/dl
HbA1c | Baseline
  percentage (%)

CONTACTS AND LOCATIONS:
Overall Officials: Lisse Angarita, PhD, Principal Investigator — Universidad Andrés Bello, Facultad de Medicina - Sede Concepción

IPD SHARING:
Plan to Share IPD: No